CLINICAL TRIAL: NCT03262922
Title: Clinical and Paraclinical Characteristics of the Systemic Scleroderma Cohort According to the Criteria ACR 2013 and the History of Professional Exposure or of Agricultural Environment
Acronym: PRESSY
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3032_PRESSY
Record Dates: First submitted 2017-08-21; First posted 2017-08-25 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Systemic Scleroderma
Keywords: systemic scleroderma; environmental and professional toxics
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to compare the exposure to environmental and professional toxics by patients with systemic scleroderma and by patients not achieved by this pathology.

DETAILED DESCRIPTION:
This study is based on a questionnaire.

The data will be collected according a retrospective and prospective design :

* at diagnostic of the disease
* at the inclusion in the systemic scleroderma cohort
* during the annual visit (in 2017-2018-2019-2020)

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic scleroderma

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic scleroderma
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Questionnaire to evaluate the exposition of environmental and professional toxics | once a year up to 2020
  clinical, personal and professional data

CONTACTS AND LOCATIONS:
Overall Officials: Patrick JEGO, Pr, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France